CLINICAL TRIAL: NCT07260435
Title: Apa/Enza Short Study: Shortened 12 Months Duration of Androgen Receptor Signaling Agent in Combination With Androgen Deprivation Therapy in Patients With Low Volume Castration-sensitive Prostate Cancer: a Randomized Nationwide Study
Brief Title: Apa/Enza-short Study: Shorter Treatment With Androgen Receptor Pathway Inhibitor in Patients With Low-volume Metastatic Castration-sensitive Prostate Cancer
Acronym: Apa/Enza-short
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nick Beije (Other)
Collaborators: Stichting Treatmeds (Unknown)
Responsible Party: Sponsor-Investigator, Nick Beije, Principal Investigator, MD PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EU CT 2023-506698-36
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADT plus continued ARPI (apalutamide/enzalutamide) (Experimental)
  Interventions: Drug: ADT plus continued ARPI
- ADT plus only 12 months of ARPI (apalutamide/enzalutamide) with the possibility t (Experimental)
  Interventions: Drug: ADT plus only 12 months of ARPI

INTERVENTIONS:
Drug: ADT plus only 12 months of ARPI — ADT plus only 12 months of ARPI (apalutamide/enzalutamide) with the possibility to resume treatment with ARSI in case of a confirmed PSA rise.
  Arms: ADT plus only 12 months of ARPI (apalutamide/enzalutamide) with the possibility t
Drug: ADT plus continued ARPI — ADT plus continued ARPI (apalutamide/enzalutamide) to the moment of progression
  Arms: ADT plus continued ARPI (apalutamide/enzalutamide)

SUMMARY:
The goal of this clinical trial is to evaluate the outcomes of a shorter treatment duration (12 months) with an androgen receptor pathway inhibitor (ARPI), in this study Apalutamide or Enzalutamide, in patients with low-volume, hormone-sensitive metastatic prostate cancer (mCSPC), with the possibility to restart treatment if needed.

The main research question is whether discontinuation of ARPI therapy after 12 months, with the option to restart treatment upon disease progression, is non-inferior to continued ARPI therapy, potentially reducing toxicity and costs.

Eligible patients will be randomized after completing 12 months of ARPI treatment, to one of the following two arms:

1. ADT + continued ARPI (Apalutamide or Enzalutamide)
2. ADT + ARPI discontinued after 12 months, with the option to resume ARPI in case of a confirmed PSA rise. The confirmatory PSA sample must be obtained at least 4 weeks after the initial rise.

This study aims to minimize toxicity associated with prolonged use of ARPIs in patients with low-volume, hormone-sensitive metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and ≥18 years of age
* Capable of understanding and complying with protocol requirements and able to understand and sign the informed consent form
* Histological diagnosis of prostate adenocarcinoma
* Low volume de novo metastatic disease (M1a or M1b) defined as anything other than fitting the criteria for high-volume metastatic disease, e.g., four or more bone lesions with one or more lesions in any body structure beyond the spine or pelvis, or visceral disease (non-nodal). This has been assessed by either bone scan and computed tomography (CT), or PSMA-PET scan. Low-volume disease has subsequently been confirmed by the local (multidisciplinary) team after consideration of the available imaging results as per the standard imaging protocol for the site.
* ADT initiated within 6 weeks prior to inclusion
* Eastern Cooperative Oncology Group (ECOG) performance scale status of 0, 1 or 2
* Fit for treatment with apalutamide or enzalutamide according to treating physician

Exclusion Criteria:

* Pathological finding consistent with small cell, ductal or neuroendocrine carcinoma of the prostate
* Other prior malignancy less than or equal to 5 years prior to randomization except for squamous or basal cell skin carcinoma or non-invasive superficial bladder cancer
* History of seizures or medications known to lower seizure threshold
* Any other prior treatment for prostate cancer other than ADT (e.g., other next generation anti-androgens or other CYP17 inhibitors, chemotherapy, immunotherapy, or radiopharmaceutical agents)
* ADT started more than 6 weeks before inclusion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to clinical progression free survival (cPFS) in both arms. | From inclusion to the last day of treatment or moment of progression (whichever occurs first). Subjects will participate for 5 years, after randomization. In total, patients will participate for 6 years.
  To prospectively evaluate whether shortened (12 months) treatment with ARPIs, with retreatment with ARPIs in case of PSA progression (defined according to PSA progression criteria) is non-inferior with respect to clinical progression free survival (boundary of max -10% at 48 months) to continued treatment with ARPI evaluated by comparing time to cPFS (as defined in primary endpoint) in both arms.

CONTACTS AND LOCATIONS:
Locations (26):
- Netherlands (26):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander MC Amersfoort, Amersfoort
  - Amsterdam Universitair Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Wilhelmina Ziekenhuis Assen, Assen
  - Rode Kruis Ziekenhuis, Beverwijk
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Treant Zorggroep, Emmen
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter ziekenhuis, Goes
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Gasthuis, Haarlem
  - Ziekenhuisgroep Twente, Hengelo
  - Tergooi MC, Hilversum
  - Frisius MC Leeuwarden, Leeuwarden
  - Maastricht UMC, Maastricht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Laurentius Ziekenhuis, Roermond
  - Bravis Ziekenhuis, Roosendaal
  - Erasmus mc, Rotterdam
  - Fransicus Gasthuis & Vlietland, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - HagaZiekenhuis, The Hague
  - St. Antonius Ziekenhuis, Utrecht
  - VieCuri Medisch Centrum, Venlo

REFERENCES:
- [Background] Stockler MR, Martin AJ, Davis ID, Dhillon HM, Begbie SD, Chi KN, Chowdhury S, Coskinas X, Frydenberg M, Hague WE, Horvath LG, Joshua AM, Lawrence NJ, Marx GM, McCaffrey J, McDermott R, McJannett M, North SA, Parnis F, Parulekar WR, Pook DW, Reaume MN, Sandhu S, Tan A, Tan TH, Thomson A, Vera-Badillo F, Williams SG, Winter DG, Yip S, Zhang AY, Zielinski RR, Sweeney CJ; ENZAMET Trial Investigators and the Australian and New Zealand Urogenital and Prostate Cancer Trials Group (ANZUP). Health-Related Quality of Life in Metastatic, Hormone-Sensitive Prostate Cancer: ENZAMET (ANZUP 1304), an International, Randomized Phase III Trial Led by ANZUP. J Clin Oncol. 2022 Mar 10;40(8):837-846. doi: 10.1200/JCO.21.00941. Epub 2021 Dec 20. PMID 34928708
- [Background] Belic J, Koch M, Ulz P, Auer M, Gerhalter T, Mohan S, Fischereder K, Petru E, Bauernhofer T, Geigl JB, Speicher MR, Heitzer E. Rapid Identification of Plasma DNA Samples with Increased ctDNA Levels by a Modified FAST-SeqS Approach. Clin Chem. 2015 Jun;61(6):838-49. doi: 10.1373/clinchem.2014.234286. Epub 2015 Apr 20. PMID 25896989
- [Background] Angus L, Deger T, Jager A, Martens JWM, de Weerd V, van Heuvel I, van den Bent MJ, Sillevis Smitt PAE, Kros JM, Bindels EMJ, Heitzer E, Sleijfer S, Jongen JLM, Wilting SM. Detection of Aneuploidy in Cerebrospinal Fluid from Patients with Breast Cancer Can Improve Diagnosis of Leptomeningeal Metastases. Clin Cancer Res. 2021 May 15;27(10):2798-2806. doi: 10.1158/1078-0432.CCR-20-3954. Epub 2021 Jan 29. PMID 33514525
- [Background] Mendelaar PAJ, Robbrecht DGJ, Rijnders M, de Wit R, de Weerd V, Deger T, Westgeest HM, Aarts MJB, Voortman J, Martens JWM, van der Veldt AAM, Nakauma-Gonzalez JA, Wilting SM, Lolkema M. Genome-wide aneuploidy detected by mFast-SeqS in circulating cell-free DNA is associated with poor response to pembrolizumab in patients with advanced urothelial cancer. Mol Oncol. 2022 May;16(10):2086-2097. doi: 10.1002/1878-0261.13196. Epub 2022 Mar 17. PMID 35181986
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Vandekerkhove G, Struss WJ, Annala M, Kallio HML, Khalaf D, Warner EW, Herberts C, Ritch E, Beja K, Loktionova Y, Hurtado-Coll A, Fazli L, So A, Black PC, Nykter M, Tammela T, Chi KN, Gleave ME, Wyatt AW. Circulating Tumor DNA Abundance and Potential Utility in De Novo Metastatic Prostate Cancer. Eur Urol. 2019 Apr;75(4):667-675. doi: 10.1016/j.eururo.2018.12.042. Epub 2019 Jan 10. PMID 30638634
- [Background] Evans CP, Higano CS, Keane T, Andriole G, Saad F, Iversen P, Miller K, Kim CS, Kimura G, Armstrong AJ, Sternberg CN, Loriot Y, de Bono J, Noonberg SB, Mansbach H, Bhattacharya S, Perabo F, Beer TM, Tombal B. The PREVAIL Study: Primary Outcomes by Site and Extent of Baseline Disease for Enzalutamide-treated Men with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer. Eur Urol. 2016 Oct;70(4):675-683. doi: 10.1016/j.eururo.2016.03.017. Epub 2016 Mar 19. PMID 27006332
- [Background] Nadal R, Taplin ME, Bellmunt J. Enzalutamide for the treatment of prostate cancer: results and implications of the AFFIRM trial. Future Oncol. 2014 Feb;10(3):351-62. doi: 10.2217/fon.13.275. PMID 24559444
- [Background] Sternberg CN, Fizazi K, Saad F, Shore ND, De Giorgi U, Penson DF, Ferreira U, Efstathiou E, Madziarska K, Kolinsky MP, Cubero DIG, Noerby B, Zohren F, Lin X, Modelska K, Sugg J, Steinberg J, Hussain M; PROSPER Investigators. Enzalutamide and Survival in Nonmetastatic, Castration-Resistant Prostate Cancer. N Engl J Med. 2020 Jun 4;382(23):2197-2206. doi: 10.1056/NEJMoa2003892. Epub 2020 May 29. PMID 32469184
- [Background] Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, Olmos D, Mainwaring PN, Lee JY, Uemura H, Lopez-Gitlitz A, Trudel GC, Espina BM, Shu Y, Park YC, Rackoff WR, Yu MK, Small EJ; SPARTAN Investigators. Apalutamide Treatment and Metastasis-free Survival in Prostate Cancer. N Engl J Med. 2018 Apr 12;378(15):1408-1418. doi: 10.1056/NEJMoa1715546. Epub 2018 Feb 8. PMID 29420164
- [Background] Hussain M, Tangen CM, Berry DL, Higano CS, Crawford ED, Liu G, Wilding G, Prescott S, Kanaga Sundaram S, Small EJ, Dawson NA, Donnelly BJ, Venner PM, Vaishampayan UN, Schellhammer PF, Quinn DI, Raghavan D, Ely B, Moinpour CM, Vogelzang NJ, Thompson IM Jr. Intermittent versus continuous androgen deprivation in prostate cancer. N Engl J Med. 2013 Apr 4;368(14):1314-25. doi: 10.1056/NEJMoa1212299. PMID 23550669
- [Background] Zhang J, Cunningham JJ, Brown JS, Gatenby RA. Integrating evolutionary dynamics into treatment of metastatic castrate-resistant prostate cancer. Nat Commun. 2017 Nov 28;8(1):1816. doi: 10.1038/s41467-017-01968-5. PMID 29180633
- [Background] James ND, de Bono JS, Spears MR, Clarke NW, Mason MD, Dearnaley DP, Ritchie AWS, Amos CL, Gilson C, Jones RJ, Matheson D, Millman R, Attard G, Chowdhury S, Cross WR, Gillessen S, Parker CC, Russell JM, Berthold DR, Brawley C, Adab F, Aung S, Birtle AJ, Bowen J, Brock S, Chakraborti P, Ferguson C, Gale J, Gray E, Hingorani M, Hoskin PJ, Lester JF, Malik ZI, McKinna F, McPhail N, Money-Kyrle J, O'Sullivan J, Parikh O, Protheroe A, Robinson A, Srihari NN, Thomas C, Wagstaff J, Wylie J, Zarkar A, Parmar MKB, Sydes MR; STAMPEDE Investigators. Abiraterone for Prostate Cancer Not Previously Treated with Hormone Therapy. N Engl J Med. 2017 Jul 27;377(4):338-351. doi: 10.1056/NEJMoa1702900. Epub 2017 Jun 3. PMID 28578639
- [Background] Chi KN, Agarwal N, Bjartell A, Chung BH, Pereira de Santana Gomes AJ, Given R, Juarez Soto A, Merseburger AS, Ozguroglu M, Uemura H, Ye D, Deprince K, Naini V, Li J, Cheng S, Yu MK, Zhang K, Larsen JS, McCarthy S, Chowdhury S; TITAN Investigators. Apalutamide for Metastatic, Castration-Sensitive Prostate Cancer. N Engl J Med. 2019 Jul 4;381(1):13-24. doi: 10.1056/NEJMoa1903307. Epub 2019 May 31. PMID 31150574
- [Background] James ND, Sydes MR, Clarke NW, Mason MD, Dearnaley DP, Spears MR, Ritchie AW, Parker CC, Russell JM, Attard G, de Bono J, Cross W, Jones RJ, Thalmann G, Amos C, Matheson D, Millman R, Alzouebi M, Beesley S, Birtle AJ, Brock S, Cathomas R, Chakraborti P, Chowdhury S, Cook A, Elliott T, Gale J, Gibbs S, Graham JD, Hetherington J, Hughes R, Laing R, McKinna F, McLaren DB, O'Sullivan JM, Parikh O, Peedell C, Protheroe A, Robinson AJ, Srihari N, Srinivasan R, Staffurth J, Sundar S, Tolan S, Tsang D, Wagstaff J, Parmar MK; STAMPEDE investigators. Addition of docetaxel, zoledronic acid, or both to first-line long-term hormone therapy in prostate cancer (STAMPEDE): survival results from an adaptive, multiarm, multistage, platform randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1163-77. doi: 10.1016/S0140-6736(15)01037-5. Epub 2015 Dec 21. PMID 26719232
- [Background] Kyriakopoulos CE, Chen YH, Carducci MA, Liu G, Jarrard DF, Hahn NM, Shevrin DH, Dreicer R, Hussain M, Eisenberger M, Kohli M, Plimack ER, Vogelzang NJ, Picus J, Cooney MM, Garcia JA, DiPaola RS, Sweeney CJ. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer: Long-Term Survival Analysis of the Randomized Phase III E3805 CHAARTED Trial. J Clin Oncol. 2018 Apr 10;36(11):1080-1087. doi: 10.1200/JCO.2017.75.3657. Epub 2018 Jan 31. PMID 29384722
- See also: Related Info — https://www.iknl.nl/kankersoorten/prostaatkanker/registratie/prevalentie